CLINICAL TRIAL: NCT06245499
Title: The Aging Brain Care Virtual Program
Brief Title: Aging Brain Care Virtual Program
Acronym: ABCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Regenstrief Institute, Inc. (Other); Indiana University Health (Other)
Responsible Party: Principal Investigator, Alexia M. Torke, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FY23_Demo2_Torke; 20249 (Other: Indiana University Institutional Review Board); U54AG063546 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Telehealth; Virtual intervention; Aging brain care
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Care Partners in the intervention group will be approached and offered care coordination through the Aging Brain Care Virtual program
  Interventions: Behavioral: Aging Brain Care Virtual Program
- Control (No Intervention): Care partners in the control group will not be approached, but outcomes data will be collected from the EMR for comparison with the intervention group.

INTERVENTIONS:
Behavioral: Aging Brain Care Virtual Program — The program involves a virtual intervention to be delivered by RN or SW care coordinators over one year. Every care partner will receive monthly virtual visits during the first 3 months and then quarterly or more depending on assessed need. The intervention relies on a tailored approach in which patient and caregiver needs are identified during visits using validated assessment tools and addressed with standardized protocols. Protocols include management of behavioral/psychological symptoms of dementia, caregiver stress, medication management, comorbidity management and advance care planning.
  Other Names: ABCV
  Arms: Intervention

SUMMARY:
The program involves a virtual intervention to be delivered by RN or SW care coordinators over one year. Every care partner will receive monthly virtual visits during the first 3 months and then quarterly or more depending on assessed need. The intervention relies on a tailored approach in which patient and caregiver needs are identified during visits using validated assessment tools and addressed with standardized protocols. Protocols include management of behavioral/psychological symptoms of dementia, caregiver stress, medication management, comorbidity management and advance care planning.

ELIGIBILITY:
Patient Inclusion Criteria:

* 65 and older,
* active primary care patient (visit in past 14 months),
* diagnosis of Alzheimer's disease and related dementias (ADRD) based on ICD criteria in primary care problems list.

Patient Exclusion Criteria:

* enrolled in hospice at the study start (study screening)or
* living in a long term care nursing facility.

Care Partners Inclusion Criteria:

* 18 and older,
* able to access a phone or computer for intervention delivery in English, and
* identified in the EMR as the emergency contact or as the primary care partner.

Care Partners Exclusion Criteria:

- Individuals who decline to participate in the ABCV intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 989 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Emergency Department Utilization | During the 12 months of intervention
  Total count of emergency department encounters per patient

SECONDARY OUTCOMES:
New prescriptions for antipsychotic medications | During the 12 months of intervention
  Total count of new prescriptions for antipsychotic medications
New prescriptions for benzodiazepine medications | During the 12 months of intervention
  Total count of new prescriptions for benzodiazepine medications
Anticholinergic Cognitive Burden Scale score | Before and 12 months after initial intervention
  Total score rating the anticholinergic burden of medications the patient is taking There are 88 medications on the Anticholinergic Cognitive Burden Scale.
  Possible anticholinergics include those listed with a score of 1; Definite anticholinergics include those listed with a score of 2 or 3.
  The overall ACB score is calculated by adding the score for each possible or definite anticholinergic medication that the patient is taking.
  An ACB Scale score can be as low as 0. The vast majority of patients have an ACB score at or below 4. Scores of 1 are low, 2 are moderate and anything above 3 is considered high. There is no published max score on the ACB scale, however, scores above 4 are somewhat uncommon. The top score could be as high as 264 (88x3)
  A higher ACB score indicates higher cognitive burden. Higher scores indicate worse outcomes.
Acceptability of the intervention score | During the 12 month intervention period
  Acceptability of Intervention Measure (AIM) Scores range from 4 to 20. Cut-off scores for interpretation are not yet available however higher scores indicate superior psychometric quality.
Feasibility of the intervention score | During the 12 month intervention period
  Feasibility of Intervention Measure (FIM) Scores range from 4 to 20. Cut-off scores for interpretation are not yet available however higher scores indicate superior psychometric quality.
Appropriateness of the intervention score | During the 12 month intervention period
  Intervention Appropriateness Measure (IAM) Scores range from 4 to 20. Cut-off scores for interpretation are not yet available however higher scores indicate superior psychometric quality.

CONTACTS AND LOCATIONS:
Overall Officials: Alexia M Torke, MD, MS, Principal Investigator — Regenstrief Institute, Inc.
Locations (1):
- Regenstrief Institute, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sauerteig-Rolston MR, Fowler NR, Sachs GA, Boustani M, Slaven J, Monahan PO, Burke ES, Higbie A, Torke AM. Pragmatic trial of a virtual dementia collaborative care management program: protocol for the Aging Brain Care Virtual (ABCV) program. BMJ Open. 2025 Sep 23;15(9):e108800. doi: 10.1136/bmjopen-2025-108800. PMID 40987722